CLINICAL TRIAL: NCT05192304
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of Multiple Doses of TPN672 Tablets Maleate in Patients With Schizophrenia
Brief Title: Evaluate the Safety, Tolerability and Pharmacokinetic Profile of TPN672 Tablets Maleate in Patients With Schizophrenia
Acronym: TPN672
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BR-2020-1491-TPN672
Record Dates: First submitted 2021-08-28; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-10

CONDITIONS: Schizophrenia
Keywords: Phase Ib; CHINA
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 0.2mg single dose (Experimental): single dose of TPN-672 0.2mg, 2 subjects
  Interventions: Drug: TPN-672
- 0.3mg single dose (Experimental): single dose of TPN-672 0.3mg, 12 subjects（9 for TPN-672, 3 for placebo）
  Interventions: Drug: TPN-672
- 0.4mg single dose (Experimental): single dose of TPN-672 0.4mg, 12 subjects（9 for TPN-672, 3 for placebo）
  Interventions: Drug: TPN-672
- 0.5mg single dose (Experimental): single dose of TPN-672 0.5mg, 12 subjects（9 for TPN-672, 3 for placebo）
  Interventions: Drug: TPN-672
- 0.6mg single dose (Experimental): single dose of TPN-672 0.6mg, 12 subjects（9 for TPN-672, 3 for placebo）
  Interventions: Drug: TPN-672
- 0.7mg single dose (Experimental): single dose of TPN-672 0.7mg, 12 subjects（9 for TPN-672, 3 for placebo）
  Interventions: Drug: TPN-672

INTERVENTIONS:
Drug: TPN-672 — single dose of TPN-672 maleate tablet
  Other Names: single dose of TPN-672 maleate tablet

SUMMARY:
This is a Phase Ib clinical study of TPN672 maleate in patients with schizophrenia

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled, dosion-increasing, Phase Ib clinical study evaluating the safety, tolerability, and pharmacokinetic characteristics of multiple doses of TPN672 maleate in patients with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 65 years old at the time of signing the informed consent form, male or female.
2. 18.5kg/m2 ≤ body mass index (BMI) ≤ 30kg/m2, and weight ≥ 50kg for men and ≥ 45kg for women.
3. Subjects met DSM-5 diagnostic criteria for a confirmed diagnosis of schizophrenia and were stable within the past 6 months as assessed by the investigator.
4. Subjects are currently taking aripiprazole, olanzapine or risperidone monotherapy for schizophrenia at a dose not exceeding the maximum dose specified in the instructions and the dose and frequency of administration have not changed in the last 1 month.
5. Screening period PANSS scale total score <70, PANSS scale individual score of positive symptom items ≤3, CGI-S score ≤4.
6. Individual scores were ≤1 on the SAS scale, ≤2 on the AIMS scale, and ≤2 on item 4 of the BARS scale, "Overall clinical assessment of sedentary inability" during the screening period.
7. Female and male subjects of childbearing potential and their spouses must be able to secure effective contraception (medically approved contraception such as IUDs, the pill or condoms) during the study and for 6 months after the end of the drug administration.
8. Subjects and their guardians fully understand the purpose and requirements of the trial, voluntarily participate in the clinical trial and sign a written informed consent form, and are willing to complete the entire trial process according to the trial requirements.

Exclusion Criteria:

1. Subjects met DSM-5 criteria for other psychiatric disorders.
2. Subjects were administered strong inducers/strong inhibitors of CYP2D6, CYP3A4, CYP3A5, CYP2C9 for 5 half-lives prior to the first dose.
3. Subjects were on long-acting antipsychotics for 6 months prior to their first dose.
4. Received electroconvulsive therapy, transcranial magnetic stimulation (rTMS) within 1 month prior to screening
5. Those who answered "yes" to questions 4 or 5 of the suicidal ideation entry on the Columbia Suicide Scale (C-SSRS) during the screening period, or who were currently or within the past 12 months significantly suicidal, or who were considered to be at risk for suicidal and violent behavior based on the investigator's clinical assessment.
6. Those with abnormal physical examination or vital signs during the screening period that are clinically significant.
7. Abnormal laboratory tests during the screening period that the investigator determines to be clinically significant, e.g., liver: ALT or AST≥ 1.2 times the upper limit of normal; kidney: Cr> the upper limit of normal value.
8. Prolactin ≥ 5 times the upper limit of normal during the screening period.
9. Screening subjects with systolic blood pressure <90 mmHg or >140 mmHg and diastolic blood pressure < 60mmHg or >90mmHg.
10. Patients with poorly controlled diabetes (fasting glucose ≥ 10 mmol/L), or are On insulin for diabetes, or at screening with a primary diagnosis of type 2 diabetes.
11. Screening QTc interval >450ms (men) or 470ms (women), or family history of long QT interval syndrome, or combined cardiac insufficiency, severe arrhythmia or ischemic heart disease requiring medication, congenital heart disease, severe organic heart disease or history of such disease.
12. Combined with convulsive disorders such as epilepsy (except febrile convulsions)
13. Current or previous hyper- or hypothyroidism, Parkinson's disease, malignancy.
14. Tobacco addiction within 1 year prior to screening, with an average of >10 cigarettes or equivalent per day.
15. Alcohol consumption within 1 year prior to screening, with an average weekly intake of more than 14 units of alcohol (1 unit = 285 ml of beer or 25 ml of spirits or 150 ml of wine) or a positive breath test for alcohol.
16. Persons with a history of drug or substance abuse within 1 year prior to screening or a positive urine drug screen.
17. Subjects who may be hypersensitive to any of the components of this drug.
18. HIV antibody, HBsAg, HCV antibody or positive syphilis serology results.
19. History of significant blood loss or blood loss ≥ 200 ml in the 3 months prior to screening
20. Enrolled in another clinical trial within 3 months prior to screening, or currently participating in a clinical trial.
21. Women who are expecting or breastfeeding.
22. The investigator did not consider it appropriate to participate in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 62 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | follow-up visit from the beginning of the dose to the day 14 after the last dose
  Incidence of Adverse Events
Blood pressure | Day 14
  Safety indicator,Blood pressure is recorded in millimeters of mercury
Respiration | Day 14
  Safety indicator，the unit of recording is the number of breaths per minute.
Heart rate | Day 14
  Safety indicator，the unit of heart rate is the number of heartbeats per minute.
Temperature | Day 14
  Safety indicator,Body temperature is recorded in degrees Celsius

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 240 hours
  Blood will be drawn from adult subjects pre-drug application and at 30min, 60min, 90min, 120min, 180min, 240min (4h), 480min (8h），720min (12h)，1440min(24h).
Time to maximum plasma concentration (Tmax) | 240 hours
  Biological sample including blood for PK will be collected at the same time point.
Area under the curve (AUC) | 240 hours
  Biological sample including blood for PK will be collected at the same time point.
steady state minimal concentration（Css_min） | 240hours
  Biological sample including blood for PK will be collected at the same time point
Elimination half-life (t1/2) | 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours ,days 8-14 after the last dose.
  Biological sample including blood for PK will be collected at the same time point.
Positive and Negative Syndrome Scale | Follow-up visit on the day 14 after the last dose
  The PANSS consisted of a positive scale of 7 items, a negative scale of 7 items, and a general psychopathology scale of 16 items, for a total of 30 items, and 3 supplementary items to assess the risk of attack. A 7-point scale with increasing levels of psychopathology was used: 1 nothing; 7 a very severe.
Clinical Global Impression sions scale | Follow-up visit on the day 14 after the last dose
  The scale is divided into 1. overall assessment of disease severity 2. overall degree of improvement. The lower the score, the higher the degree of improvement of the patient.
Calgary Depression Scale for Schizophrenia | Follow-up visit on the day 14 after the last dose
  There were 9 entries, including mood depression, feelings of hopelessness, self-deprecation, guilt implicated perceptions, pathological guilt, morning depression, early awakening, suicidality, and observed depressive manifestations. The lower the score the less severe the depressive symptoms.
Blood coagulation function | Day 14
  Safety indicators, including PT,APTT
12-lead ECG | Day 14
  Safety indicators, including QTc
Serum prolactin ( PRL) | Day 14
  Testing for affected hormone levels

CONTACTS AND LOCATIONS:
Overall Officials: Li Huafang, MD PhD, Principal Investigator — Shanghai Mental Health Center; Li Guanjun, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No